CLINICAL TRIAL: NCT03949023
Title: Influence of Contrast Injection Force on the Accuracy of Vessel Measurements in Cerebral Angiography
Status: Terminated | Type: Observational
Why Stopped: unable to perform refinement of study procedures to better capture information needed
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00049517
Record Dates: First submitted 2019-05-07; First posted 2019-05-14 (Actual); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: Cerebral Angiogram
Keywords: Neurovascular Condition; Contrast Injections; Brain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Standard of Care Cerebral Angiogram Group: Participants undergoing a standard of care cerebral angiogram.
  Interventions: Procedure: Standard of Care Cerebral Angiogram Group

INTERVENTIONS:
Procedure: Standard of Care Cerebral Angiogram Group — Subjects will undergo the standard of care cerebral angiogram and any intervention(s) (when applicable) that were discussed with their provider, following the standard procedural protocol for the procedure at WFBMC. There are no additional interventions or changes to the planned intervention(s) that will take place by agreeing to participate in the study.
  The data collected from this procedure, following the standard of care protocol, will include the following: force of injection of contrast material for each angiographic run (peak pressure associated with injection, duration of peak, and area under pressure curve), volume of contrast utilized, images from the procedure, measurements of vessel diameter at defined distances from the catheter tip utilizing the images, catheter type, any additional device(s) (when applicable) utilized during the procedure, and if spasmolytic agents are utilized (including dose and time of administration).

SUMMARY:
The purpose of this research study is to collect data/measurements that are routinely collected in standard of care cerebral angiogram

DETAILED DESCRIPTION:
Research for this study is to determine how the injection of contrast material influences vessel measurements, as these measurements guide device selection when interventions are warranted.

The data will be used to determine if there is a significant change in vessel diameter with intra-arterial injection of contrast material in cerebral angiography, how changes in force of contrast injection augments the significance of the changes in vessel geometry, and the extent of propagation downstream from the catheter tip that such changes in vessel diameter are detected and found to be significant, as these changes could potentially lead to less optimal device selection by providing an overestimation of true vessel diameter.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving care at WFBMC that will be undergoing a standard of care cerebral angiogram who are anticipated to have a minimum of 2 images for an individual view required for the necessary data collection

Exclusion Criteria:

* Patients who are anticipated to have less than 2 images for each standard view collected from their cerebral angiogram.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving care at WFBMC that will be undergoing a standard of care cerebral angiogram that are anticipated to have multiple images per standard view (a minimum of 2 images for an individual view required for the necessary data collection).
  Patients that are anticipated to have less than 2 images for each standard view collected from their cerebral angiogram.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2018-07-12 (Actual); Primary Completion 2018-07-12 (Actual); Study Completion 2018-07-12 (Actual)

PRIMARY OUTCOMES:
Peak pressure associated with injection | During procedure, up to 10 minutes
  The effort force of injection will be measured and recorded for each run using a standard arterial line pressure transducer setup that attaches to the guide catheter, with data acquired via Mediocollector (a program that allows for quantitative recording of data. The duration of peak pressure will be collected.
The duration of peak pressure | During procedure, up to 10 minutes
  The duration of peak pressure will be collected.

OTHER OUTCOMES:
Vessel Diameter | During the procedure, up to 10 minutes
  Measurement of vessel diameter

CONTACTS AND LOCATIONS:
Overall Officials: Kyle M Fargen, MD, Ph.D, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] S P Sutera a, Skalak R. The History of Poiseuille's Law. Annual Review of Fluid Mechanics. 1993;25(1):1-20
- [Background] Yousem DM, Trinh BC. Injection rates for neuroangiography: results of a survey. AJNR Am J Neuroradiol. 2001 Nov-Dec;22(10):1838-40. PMID 11733311
- [Background] Hao Q, Lieber BB. Dispersive Transport of Angiographic Contrast During Antegrade Arterial Injection. Cardiovasc Eng Technol. 2012 Jun 1;3(2):171-178. doi: 10.1007/s13239-012-0090-x. Epub 2012 Apr 13. PMID 23139732
- [Background] Alexander MD, Nicholson AD, Darflinger RJ, Settecase F, Cooke DL, Dowd CF, Amans MR, Higashida RT, Hetts SW, Halbach VV. Effects on vessel measurement accuracy and subsequent occlusion after calcium channel blocker infusion during treatment of cerebral aneurysms with the Pipeline embolization device. Interv Neuroradiol. 2017 Feb;23(1):47-51. doi: 10.1177/1591019916674916. Epub 2016 Oct 27. PMID 27798327